CLINICAL TRIAL: NCT06725992
Title: A Randomized, Open-label, Multiple-dose, Crossover Phase 1 Clinical Trial to Compare and Evaluate the Safety, PK and PD Characteristics After Oral Administration of IY-NS250 and IY-NT-SR in Healthy Adult Volunteers
Brief Title: Study to Evaluate Pharmacokinetic and Pharmacodynamic Drug Interactions and Safety of IY-NS250 and IY-NT-SR
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Il-Yang Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IY-NS250SB
Record Dates: First submitted 2024-02-21; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Pharmacokinetics; Pharmacodynamics

STUDY DESIGN:
Intervention Model Description: A randomized, open-label, multiple-dose, crossover phase 1 clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A group (Active Comparator): Period 1 : Ilaprazole 10mg 2Tab, one a day
  Period 2 : IY-NS250 1Tab, one a day
  Interventions: Drug: IY-NS250; Drug: IY-NT-SR
- B group (Active Comparator): Period 1 : IY-NS250 1Tab, one a day
  Period 2 : Ilaprazole 10mg 2Tab, one a day
  Interventions: Drug: IY-NS250; Drug: IY-NT-SR

INTERVENTIONS:
Drug: IY-NS250 — Ilaprazole 20mg + Sodium bicarbonate 500mg
Drug: IY-NT-SR — Ilaprazole 10mg
  Other Names: Noltec(the brand name)

SUMMARY:
This study comparative evaluation of safety and pharmacokinetic and pharmacodynamic properties in oral repeat administration of IY-NS250 and IY-NT-SR in healthy adult

DETAILED DESCRIPTION:
Not provided

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult volunteers aged 19 years or older at screening
2. Individuals with a weight of 50.0 kg or more and a body mass index (BMI) of 18.0 kg/m2 to 30.0 kg/m2 at screening

   * BMI (kg/m2) = Weight (kg) / {Height (m)}2
3. ndividuals without congenital or chronic diseases requiring treatment and with no pathological symptoms or findings from internal medical examinations (if necessary, brain waves, electrocardiograms, chest and upper gastrointestinal endoscopy or gastrointestinal radiographic examinations)
4. Individuals deemed suitable for the clinical trial based on clinical trial laboratory tests, vitality signs, physical examinations, and 12-lead electrocardiogram results conducted according to the characteristics of the investigational product at screening
5. Individuals with negative H. pylori antibody results at screening
6. Individuals who have heard a detailed explanation of the clinical trial, fully understand it, voluntarily decide to participate, and agree in writing to comply with the subject compliance requirements during the clinical trial period

Exclusion Criteria:

1. Individuals with a current or past medical history of clinically significant conditions affecting the liver, kidneys, nervous system, psychiatric system, respiratory system, endocrine system, hematologic disorders, tumors, genitourinary system, cardiovascular system, digestive system, musculoskeletal system, or any of the following current or past conditions:

   * Renal impairment

     * Hepatic impairment
2. Individuals with a history of gastrointestinal disorders (such as Crohn's disease, ulcers, acute or chronic pancreatitis) or gastrointestinal surgery (excluding simple appendectomy or hernia repair) that may affect the absorption of investigational drugs
3. Women who are pregnant (as indicated by positive Urine-HCG) or lactating
4. Individuals with a history of hypersensitivity reactions (such as anaphylaxis or angioedema) or clinically significant hypersensitivity reactions to drugs containing Ilaprazole, excipients (Tartrazine, Sunset Yellow FCF), or other drugs (such as aspirin, penicillin antibiotics, macrolide antibiotics)
5. Individuals with clinically significant findings, including the following, on the 12-lead electrocardiogram performed at screening:

   * QTc > 450 ms for males or QTc > 470 ms for females
   * PR interval > 200 ms
   * QRS duration > 120 ms
6. Individuals with clinically significant results, including the following, on clinical trial laboratory tests performed at screening:

   * AST, ALT, ALP, γ-GT, and total bilirubin levels exceeding twice the upper limit of the normal range for liver function evaluation
   * Serum creatinine levels outside the reference range or estimated glomerular filtration rate (eGFR) calculated by CKD-EPI formula < 60 mL/min/1.73m2
7. Individuals with a history of drug abuse or positive urine drug test results for abused drugs
8. Individuals with systolic blood pressure ≥ 150 mmHg or ≤ 90 mmHg, or diastolic blood pressure ≥ 100 mmHg or ≤ 60 mmHg, or heart rate ≤ 40 bpm or ≥ 100 bpm upon measurement in the supine position after resting for more than 3 minutes at screening
9. Individuals with abnormal diets that may affect the absorption, distribution, metabolism, and excretion of investigational drugs or affect drug metabolism
10. Individuals who have taken any prescription drugs or herbal medicines that may affect the characteristics of investigational drugs within 2 weeks prior to the first dosing day or any over-the-counter drugs or vitamin supplements within 10 days prior to the first dosing day (however, participation in the clinical trial may be allowed based on the participant's judgment if the drug does not affect the pharmacokinetic properties of the investigational drug)
11. Individuals who have been administered inducers or inhibitors of drug metabolism, such as barbiturates, within 1 month prior to the first dosing day
12. Individuals who have participated in another clinical trial and received treatment within 6 months prior to the first dosing day (however, the end date of participation in another clinical trial is calculated as 1 day after the last dosing day)
13. Individuals who have donated whole blood within 2 months or component blood within 1 month prior to the first dosing day, received blood transfusions within 1 month, or cannot abstain from blood donation from the time of written consent until PSV
14. Individuals who have consumed alcohol excessively (more than 21 units/week, 1 unit = 10 g = 12.5 mL of pure alcohol) within 6 months prior to the first dosing day or cannot abstain from the time of written consent until PSV
15. Individuals who have consumed grapefruit-containing foods from 48 hours before the first dosing to PSV or cannot abstain from consumption
16. Individuals who have engaged in vigorous exercise exceeding their usual daily activities from 48 hours before the first dosing to PSV or cannot abstain from such exercise
17. Individuals who, from the time of written consent until 2 weeks after the last dosing day based on the date of the last administration of investigational drugs, are not using or planning to use recognized contraceptive methods for planning or not planning pregnancy (e.g., contraceptive pills and implants, intrauterine devices, infertility procedures (vasectomy, tubal ligation), barrier methods (combined use of spermicides with condoms, vaginal sponges, cervical caps))
18. Individuals for whom insertion and maintenance of a pH meter catheter for gastric pH measurement is difficult
19. Individuals who are deemed unsuitable for participation in the clinical trial by the investigator for reasons other than the selection/exclusion criteria mentioned above.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2024-01-30 (Actual); Primary Completion 2024-04-13 (Actual); Study Completion 2024-08-14 (Actual)

PRIMARY OUTCOMES:
Ilaprazole AUCτ,ss | Day 1 Predose(0hour), after dose 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 24 hour / Day 5, Day 6 Predose(0hour) / Day 7 Predose(0hour), after dose 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 24 hour
  Ilaprazole AUCτ,ss
integrated gastric acidity | Day -1 -24hour ~ 0h Day7 Predose(0hour) ~ 24hour
  Percentage decrease in integrated gastric acidity over 24 hours from Day -1 to Day 7

SECONDARY OUTCOMES:
AUCinf,ss | Day 1 Predose(0hour), after dose 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 24 hour / Day 5, Day 6 Predose(0hour) / Day 7 Predose(0hour), after dose 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 24 hour
  AUCinf,ss, of Ilaprazole after repeated administration
Cmax,ss | Day 1 Predose(0hour), after dose 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 24 hour / Day 5, Day 6 Predose(0hour) / Day 7 Predose(0hour), after dose 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 24 hour
  Cmax,ss of Ilaprazole after repeated administration
Cmin,ss | Day 1 Predose(0hour), after dose 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 24 hour / Day 5, Day 6 Predose(0hour) / Day 7 Predose(0hour), after dose 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 24 hour
  Cmin,ss of Ilaprazole after repeated administration
Cav,ss | Day 1 Predose(0hour), after dose 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 24 hour / Day 5, Day 6 Predose(0hour) / Day 7 Predose(0hour), after dose 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 24 hour
  Cav,ss of Ilaprazole after repeated administration
Tmax,ss | Day 1 Predose(0hour), after dose 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 24 hour / Day 5, Day 6 Predose(0hour) / Day 7 Predose(0hour), after dose 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 24 hour
  Tmax,ss of Ilaprazole after repeated administration
t1/2,ss | Day 1 Predose(0hour), after dose 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 24 hour / Day 5, Day 6 Predose(0hour) / Day 7 Predose(0hour), after dose 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 24 hour
  t1/2,ss of Ilaprazole after repeated administration
CLss/F | Day 1 Predose(0hour), after dose 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 24 hour / Day 5, Day 6 Predose(0hour) / Day 7 Predose(0hour), after dose 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 24 hour
  CLss/F of Ilaprazole after repeated administration
Vss/F, R (accumulation ratio) | Day 1 Predose(0hour), after dose 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 24 hour / Day 5, Day 6 Predose(0hour) / Day 7 Predose(0hour), after dose 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 24 hour
  Vss/F, R (accumulation ratio) of Ilaprazole after repeated administration
PTF (Peak to Trough fluctuation) | Day 1 Predose(0hour), after dose 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 24 hour / Day 5, Day 6 Predose(0hour) / Day 7 Predose(0hour), after dose 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 24 hour
  PTF (Peak to Trough fluctuation) of Ilaprazole after repeated administration
Cmax | Day 1 Predose(0hour), after dose 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 24 hour
  Cmax of Ilaprazole after single administration
AUClast | Day 1 Predose(0hour), after dose 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 24 hour
  AUClast of Ilaprazole after single administration
AUCinf | Day 1 Predose(0hour), after dose 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 24 hour
  AUCinf of Ilaprazole after single administration
Tmax | Day 1 Predose(0hour), after dose 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 24 hour
  Tmax of Ilaprazole after single administration
t1/2 | Day 1 Predose(0hour), after dose 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 24 hour
  t1/2 of Ilaprazole after single administration
CL/F | Day 1 Predose(0hour), after dose 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 24 hour
  CL/F of Ilaprazole after single administration
Vz/F | Day 1 Predose(0hour), after dose 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 24 hour
  Vz/F of Ilaprazole after single administration
integrated gastric acidity | Day -1 -24hour ~ 0h Day 1 Predose(0hour) ~ 24h Day7 Predose(0hour) ~ 24hour
  Percentage decrease in integrated gastric acidity at different time points from Day -1 to Day 1 and Day 7
nocturnal acid breakthrough (NAB) | Day -1 -24hour ~ 0h Day 1 Predose(0hour) ~ 24h Day7 Predose(0hour) ~ 24hour
  Percentage of subjects experiencing nocturnal acid breakthrough (NAB) on Day -1, Day 1, and Day 7, defined as maintaining a pH below 4 for more than 60 consecutive minutes during nighttime (supine position)

CONTACTS AND LOCATIONS:
Overall Officials: Min Kyu Park, MD, PhD, Principal Investigator — Chungbuk National University Hospital
Locations (1):
- Chungbuk National University Hospital, Seoul, Seowon-gu, South Korea